CLINICAL TRIAL: NCT06238284
Title: HER2 Expression in Gynecological Malignant Tumors in Chongqing Area of China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CQ-HER2-GYN
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Cancer; HER2 Expression
Keywords: Cervical Cancer; Endometrial Cancer; Ovarian Cancer; HER2 Expression; Therapeutic efficacy; Prognosis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cervical Cancer Group
  Interventions: Other: no intervention
- Endometrial Cancer Group
  Interventions: Other: no intervention
- Ovarian Cancer Group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Since it is a retrospective study, no intervention is needed.

SUMMARY:
This study aims to retrospectively analyze the HER2 expression of gynecological malignant tumors in Chongqing by immunohistochemical detection, and explore the correlation between HER2 level, therapy response and prognosis based on patient clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary gynecological malignant tumor confirmed by histopathology
* Women aged 18-75
* The expected survival time is greater than 12 weeks
* KPS > 60, ECOG score is 0-2
* All subjects voluntarily joined this study with informed consents, and had good compliance of follow-up

Exclusion Criteria:

* Pregnant and lactating women
* Suffering from other malignant tumors in the past 5 years
* Patients who are not suitable for this study according to the investigator's judgment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with cervical adenocarcinoma (including carcinosarcoma), adenocarcinoma of uterus (including carcinosarcoma), or ovarian cancer, etc.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-26 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
HER2 status | from 2023.07 to 2024.05
  HER2 exprssion level evaluated by pathologists